CLINICAL TRIAL: NCT06666465
Title: Operating Room Environment Experienced by Patients With Virtual Reality Glasses Before Surgery The Effect of Surgical Experience on the Level of Surgical Fear and Perceptions of Care
Brief Title: The Effect of the Operating Room Environment on Patients Experienced With Virtual Reality Glasses Before Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, İmren Erer, Msc, Saglik Bilimleri Universitesi
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: ierer
Record Dates: First submitted 2024-08-23; First posted 2024-10-30 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Clinical Practice; Virtual Reality; Nursing Care; Simulation
Keywords: Clinical practice

STUDY DESIGN:
Intervention Model Description: Patients participating in the study will be included in a group by gender-based stratified block randomization method. Patients in the intervention group will experience the operating room environment with VR glasses (n: 30), while patients in the control group (n: 30) will receive standard nursing care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Operating Room Environment Experienced by Patients (Experimental): This study was planned as a randomized controlled experimental study in the pre-test post-test design in order to examine the effect of the operating room environment experience of patients using virtual reality glasses before surgery on the level of surgical fear experienced by patients before surgery and their perception of care.
  Interventions: Other: Operating Room Environment Experienced by Patients Wearing Virtual Reality Glasses Before Surgery The Effect of Surgery Experience on Surgical Fear Level and Care Perceptions

INTERVENTIONS:
Other: Operating Room Environment Experienced by Patients Wearing Virtual Reality Glasses Before Surgery The Effect of Surgery Experience on Surgical Fear Level and Care Perceptions — The video, which will be shot for patients to experience the operating environment, will include premedication, an operating room and a post-operative care unit. In the video, the operating room environment will be recorded by the researcher with a voice introduction. The image was shot with a 360-degree camera (Insta 360 One X2), edited with an application program (Insta 360 Studio) and then uploaded to the YouTube VR Pro application as a secret video. The video will be shown to the glasses via an Android phone on the internet via YouTube. People wearing glasses at the screening will be able to look in any direction they want thanks to the 360-degree video. They will be able to watch the video again if they want.

SUMMARY:
This study was planned as a randomized controlled experimental study with a pretest-posttest design to examine the effect of the operating room environment experience of preoperative patients using virtual reality glasses on the patients' preoperative surgical fear level and care perceptions.

DETAILED DESCRIPTION:
Today, virtual reality is used in many areas such as medical diagnosis and treatment by reflecting three-dimensional images animated on the computer as if it were a real experience. Procedural pain, facilitating interventional procedures with a game-based video demonstration in children, and outpatient surgeries such as circumcision surgery can be used to provide patients with this "real world" experience, its use has also become widespread in areas such as wound care and in nursing education due to the increase in malpractice cases . In line with patient experiences, the benefits of virtual reality technology have been documented in the literature and its use in nursing care is increasing . Informing the patient to improve the quality of care, managing pain during painful interventional procedures, and reducing surgery-related fear reduces wound healing and hospital stay, especially in surgical patients . In the literature, patients' pre-operative problems such as lack of knowledge about the surgery, operating room environment, surgical procedures, etc. It is reported that they experience anxiety and fear related to many factors. It also emphasizes the importance of informing the patient before surgery within the scope of Enhance Recovery After Surgery (ERAS) procedures (Joshi & Kehlet, 2019). In line with ERAS protocols, preoperative education and information have been proven to provide positive postoperative recovery. Informing the patient about the operating room environment is the most important element in accelerating surgical recovery. The operating room environment can be seen as a stress factor for patients. Therefore, in this study, we aimed to examine the effect of informing patients about the operating room environment, supported by visuals, on the patient's fear and perceptions of care. In addition, it is thought that this information and experience will affect the patient's vital signs and that the patient's need for premedication will also change. It is thought that the results of this study will positively affect patient outcomes by improving the quality of patient care.

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years or older
* Agreeing to participate in the research
* Having elective cholecystectomy surgery
* Knowledge of Turkish and no communication barriers
* Having surgery for the first time and not having seen the operating room environment

Exclusion Criteria:

* Being 18 years of age or younger
* Refusal to participate in the research
* Having undergone surgery and having seen the operating room environment before Not knowing Turkish and having any communication barrier

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — patients undergoing surgery
Enrollment: 60 (Estimated)
Dates: Start 2024-08-15 (Actual); Primary Completion 2025-12-16 (Estimated); Study Completion 2025-12-20 (Estimated)

PRIMARY OUTCOMES:
Change in surgical fear levels of patients in the operating environment after simulation experience with virtual reality glasses | Preoperative Use of Virtual Reality After Simulation
  Change in Anxiety and Stress Levels during the care of patients undergoing surgery Simulation of the operating room environment to patients using virtual reality glasses will affect patients' stress and anxiety levels in the operating room. This situation will be evaluated. The scale consists of 8 items, scored from 0 to 10, and is an 11-point Likert-type scale. Each item is scored as 0 "not at all afraid" and 10 "very afraid". The scale consists of two sub-dimensions, each consisting of four items. These indicate the fear of short-term and long-term consequences of surgery; items 1-4 in the scale measure the fear of short-term consequences of surgery, while items 5-8 measure the fear of long-term consequences of surgery.
change in patients' perceptions of nursing care | Preoperative Use of Virtual Reality After Simulation
  The change in patients' nursing care perception scores will be measured. There are 15 statements on the Likert-type scale regarding the quality of nursing care. It is requested to mark one of the 15 statements that make up the scale: I agree = 5, I somewhat agree = 4, I am undecided = 3, I disagree = 2, I strongly disagree = 1 and no response = 0. The score given for each item is taken as basis. Thus, a minimum of 15 and a maximum of 75 points can be obtained from the scale. The increase in the total score obtained from the scale indicates that the patient is satisfied with the nursing care.

CONTACTS AND LOCATIONS:
Overall Officials: Emine Parlak, 2, Study Chair — Saglik Bilimleri Universitesi
Locations (1):
- İmren Erer, İnönü, Eskişehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Addab, S., Hamdy, R., & Thorstad, K. (2022). Use of Virtual Reality in Managing Pediatric Prosedural Pain and Anxiety: an Integrative Literature Review. Journal of Clinical Nursing, 31(21-22), s. 3032-3059. Ahern, M., Dean, L., Stoddard, C., Agrawai, A., Kim, K., Cook, C., & Garcia, A. (2020). The Effectviveness of Virtual Reality in Patients with Spinal Pain: Systematic Review and Meta- Analysis. Pain Practice, 20(6), s. 656-675. Baytar, Ç., & Bollucuoğlu, K. (2021). Effect of Virtual Reality on Preoperative Anxiety Inpatients Undergoing septorhinoplasty. Brazilian Journal of Anesthesiology, 1(744276), s. 1-6. Bağdigen Kaya, M., & Karaman Özlü, Z. (2019). Elektif Cerrahi Bekleyen Hastalarda Cerrahi Korkunun Sosyal Destek Algısı ile İlişkisinin Belirlenmesi. Anadolu Hemşirelik ve Sağlık Bilimleri Dergisi, 22(4), s. 281-290.